CLINICAL TRIAL: NCT03887897
Title: A Randomized Controlled Trial to Compare the First-pass Intubation Success of the Airtraq Laryngoscope Versus the Macintosh Direct Laryngoscope in Patients Requiring General Anaesthesia for Elective Operation.
Brief Title: First Attempt Intubation Rate With Airtraq vs Macintosh Direct Laryngoscope
Acronym: FAIRAiM
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese University of Hong Kong (Other)
Collaborators: Tuen Mun Hospital (Other Government)
Responsible Party: Principal Investigator, Matthew Chan, Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: FAIR AiM protocol V1.0
Record Dates: First submitted 2019-03-20; First posted 2019-03-25 (Actual); Last update posted 2019-11-12 (Actual); Status verified 2019-11

CONDITIONS: Intubation
Keywords: First-pass; first attempt;intubation success
MeSH Terms: interventions — Intubation, Intratracheal

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Airtraq (Active Comparator): Airtraq laryngoscope
  Interventions: Procedure: Tracheal Intubation
- Macintosh (Active Comparator): Macintosh laryngoscope
  Interventions: Procedure: Tracheal Intubation

INTERVENTIONS:
Procedure: Tracheal Intubation — Tracheal intubation performed by attending anesthesiologists using either Airtraq laryngoscope or Macintosh laryngoscope

SUMMARY:
In recent decades, numerous videolaryngoscopes have been introduced to facilitate tracheal intubation. However, it remains unclear whether videolaryngoscope will increase the successful tracheal intubation compared with usual Macintosch laryngoscope. Therefore, this pilot study is a randomized controlled trial designed to compare the first-pass intubation success of the Airtraq laryngoscope versus the Macintosh direct laryngoscope in patients requiring general anesthesia for elective operation, with the aims to examine the feasibility of a large multicentre effectiveness trial by assessing recruitment targets, testing the data completeness, and local incidence of first-pass intubation success.

DETAILED DESCRIPTION:
In recent decades, numerous videolaryngoscopes have been introduced to facilitate tracheal intubation. However, it remains unclear whether videolaryngoscope will increase the successful tracheal intubation compared with usual Macintosch laryngoscope. In a quantitative review on the performance of several non-standard laryngoscopes (e.g. Bonfils, CTrach, Glidescope), no strong evidence has been identified to support these devices to supersede the Macintosh laryngoscope. Owing to the lacks of randomized trials at the time, Airtraq has not been reviewed in the analysis.

The Airtraq laryngoscope is one of the optical indirect laryngoscopes, which provides glottis display without any deviation in the normal position of the oral, pharyngeal or the tracheal axes. Unlike other videolaryngoscopes, the Airtraq larygoscope is a non-steering novel airway device which has a guide channel for tracheal tube alongside with the blade. Its use has been showed to improve the ease of intubation in difficult airway situations. Up to date, randomized controlled trials comparing the Airtraq and Macintosh direct laryngoscopes are either small scaled or focusing on specific populations. And instead of the first-attempt success rate, the primary endpoints adopted have focused on the glottic view, intubation time, and cervical spine movement. The Difficult Airway Society has highlighted the importance of a robust and high standard of evidence to assess the use of new devices in airway management. Knowing that failed tracheal intubation has remained a major contribution to anesthetic-related morbidity and mortality, clinical relevant endpoint is essential to guide the selection of airway devices for tracheal intubation. Considering reports on unsuccessful tracheal intubation under satisfactory video-laryngoscopic view, using laryngoscopic view as a surrogate measure for successful intubation can give false assurances of device efficacy. While improvement in first-pass laryngoscopic success confers less airway trauma and possibly the prevention in deterioration to a 'Cannot Intubate Cannot Ventilate' scenario, it then translates into much more success than the improvement with multiple attempts and shortened intubation time. Meta-analyses have demonstrated that the Airtraq significantly decreased intubation time both in novice and in experienced anaesthetists compared with the Macintosh laryngoscope. Whereas in the first-attempt intubation, an increase in the first-pass success rate was only found in novice anaesthetists with significant analysis heterogeneity.

In view of these, a large pragmatic effectiveness trial using first-pass intubation success as the primary endpoint to compare the Airtraq and Macinotosh direct laryngoscope is necessary. The trial population should include normal and abnormal airways, a variety of elective and non-elective patients and proceduralists with mixed experience to allow results to be generalizable. A large trial would allow testing of subgroup effects that has not been previously possible and results would be generalizable due to its pragmatic design. The results of this trial will provide improved guidance for current airway algorithms.

ELIGIBILITY:
Inclusion Criteria:

1. adult (>18years) patients;
2. receiving general anaesthesia that requires tracheal intubation

Exclusion Criteria:

1. known or predicted difficult bag-mask ventilation
2. patients scheduled for (awake or asleep) fibreoptic intubation
3. patients requiring rapid sequence intubation
4. language or congnitive problems that preclude adequate informed consent being obtained
5. patient or anaesthetist refusal.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1586 (Estimated)
Dates: Start 2019-10-02 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
First-pass success in tracheal intubation | During tracheal intubation procedure
  Successful tracheal intubation during the first attempt, confirmed by EtCO2 tracing

SECONDARY OUTCOMES:
Time to successful tracheal intubation | During tracheal intubation procedure
  Duration when laryngoscope was inserted into mouth and successful tracheal intubation with the first appearance of EtCO2 tracing
Hoarseness | At 48 hours after operation
  Subjective report of hoarseness in terms of serverity (0=nil; 1=mild; 2=moderate; 3= severe)
Sore throat | At 48 hours after operation
  Subjective report of sore throat in terms of serverity (0=nil; 1=mild; 2=moderate; 3= severe)
Use of adjuncts during tracheal intubation | During tracheal intubation procedure
  Adjuncts e.g. bougie, stylet used for tracheal intubation
Requirement of additional maneuvers | During tracheal intubation procedure
  Use of additional maneuvers applied to facilitate tracheal intubation e.g. BUPA, patient re-positioning during tracheal intubation

CONTACTS AND LOCATIONS:
Overall Officials: Mathew TV Chan, MBBS, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Department of Anaesthesia and Intensive Care, New Territories West Cluster, Hospital Authority, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mihai R, Blair E, Kay H, Cook TM. A quantitative review and meta-analysis of performance of non-standard laryngoscopes and rigid fibreoptic intubation aids. Anaesthesia. 2008 Jul;63(7):745-60. doi: 10.1111/j.1365-2044.2008.05489.x. PMID 18582261